CLINICAL TRIAL: NCT01918137
Title: A Randomised Trial of Effect of Deep-fried Chocolate Bar and Porridge Upon Cerebrovascular Reactivity in Healthy Adult Volunteers
Brief Title: The Effect of a Deep-fried Chocolate Bar or Porridge on Cerebral Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GN13MT357
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Effect on Cerebrovascular Reactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chocolate bar (Experimental)
  Interventions: Dietary Supplement: chocolate bar
- porridge (Experimental)
  Interventions: Dietary Supplement: Porridge

INTERVENTIONS:
Dietary Supplement: chocolate bar
  Arms: chocolate bar
Dietary Supplement: Porridge
  Arms: porridge

SUMMARY:
The deep fried chocolate bar is a snack that the international community strongly associates with Scotland. It has previously been cited as being "a symbol of all that is wrong with the high-fat, high-sugar Scottish diet". Despite the snack's reputation, no medical research has been performed to examine the effects of consuming a deep fried chocolate bar on the human body.

In contrast to the deep fried chocolate bar, porridge has been shown to reduce the risk of cardiovascular disease, but its effect on cerebral blood flow has yet to be directly assessed.

This study will focus on the potential (patho)physiological cerebrovascular effects of the deep fried chocolate bar and porridge. The research question to be addressed in this study is "Does eating a deep fried chocolate bar or bowl of porridge induce changes in cerebral blood flow and cereborvascular reactivity in healthy adults?"

To assess the acute effects on eating either food on blood flow through the largest artery in the brain, the investigators will give healthy volunteers one regular-sized deep-fried chocolate bar or a bowl of porridge. Blood flow through the largest artery in the brain will be assessed using simple ultrasounds tests. The investigators aim to recruit 24 volunterrs who will visit twice, consuming a different food on each visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30
* No regular medication
* Able to provide informed consent

Exclusion Criteria:

* Distaste for or contraindication to deep-fried chocolate bar or porridge ingestion
* inability to perform breath-hold

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change in breath hold index after ingestion of deep-fried chocolate bar compared with change after porridge ingestion | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Western Infirmary, Glasgow, United Kingdom